CLINICAL TRIAL: NCT02550990
Title: Synergistic Effects of Aerobic Exercise and Cognitive Training on Cognition, Physiological Markers, Daily Function and Quality of Life in Stroke Patients With Cognitive Decline
Brief Title: Synergistic Effects of Aerobic Exercise and Cognitive Training on Cognition in Stroke Patients With Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104-4892A3
Record Dates: First submitted 2015-09-06; First posted 2015-09-16 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Stroke Patients With Cognitive Decline
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive training group (Active Comparator): One 60-min session of cognitive training. Before and after the treatment, a total of 2 evaluations were conducted, including clinical assessments and blood test (each 18c.c.). A saliva sample (2 mL) will only be collected once from each subject. A follow-up assessment of clinical outcomes will be conducted at six month after the end of the course of treatment.
  Interventions: Behavioral: Cognitive training
- Aerobic exercise training group (Active Comparator): One 60-min session of aerobic exercise training. Before and after the treatment, a total of 2 evaluations were conducted, including clinical assessments and blood test (each 18c.c.). A saliva sample (2 mL) will only be collected once from each subject. A follow-up assessment of clinical outcomes will be conducted at six month after the end of the course of treatment.
  Interventions: Behavioral: Aerobic exercise training
- Sequential training group (Experimental): One 30-min session of aerobic exercise training + one 30-min session of cognitive training.
  Before and after the treatment, a total of 2 evaluations were conducted, including clinical assessments and blood test (each 18c.c.). A saliva sample (2 mL) will only be collected once from each subject. A follow-up assessment of clinical outcomes will be conducted at six month after the end of the course of treatment.
  Interventions: Behavioral: Sequential combination of aerobic exercise and cognitive training

INTERVENTIONS:
Behavioral: Cognitive training
  Arms: Cognitive training group
Behavioral: Aerobic exercise training
  Arms: Aerobic exercise training group
Behavioral: Sequential combination of aerobic exercise and cognitive training
  Arms: Sequential training group

SUMMARY:
The purpose of this study is to determine the treatment effects of sequential combination of aerobic exercise and cognitive training on cognitive function, physiological markers, daily function, physical function, social participation and quality of life in stroke patients with cognitive decline. The investigators hypothesized that: (1) sequential training protocol can improve outcome measures compared to single mode of training; (2) these treatment effects will retain at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrhagic stroke occurring at least 6 months prior to enrollment
2. Age range from 20 to 90 years
3. MMSE score ≥ 19
4. MoCA<26
5. Self- or informant-reported memory or cognitive complaints or CDR scale ≤ 0.5
6. Able to follow the study instruction
7. Adequate cardiopulmonary function to perform aerobic exercise
8. Able to walk with or without assistive devices

Exclusion Criteria:

1. Unstable medical history (e.g., recent myocardial infarction) that might limit participation
2. Concomitant with other neurological disorders (e.g., Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis)
3. Current participation in another interventional trial

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Wechsler Memory Scale - Third Edition (WMS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Useful Field of View (UFOV) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Stroop Color-Word test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Dual-task test | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  The dual-task tests will be assessed to determine the ability for an individual to perform 2 tasks simultaneously. The investigators will assess the dual-task performance during walking and performing box and block test. The results of the dual-task tests will provide information regarding to whether the 2 tasks compete for the same class of neural resources or one of the tasks can be carried out automatically.

SECONDARY OUTCOMES:
Change scores of serum BDNF level | Baseline, posttest (an expected average of 3 months)
Change scores of Antioxidative marker | Baseline, posttest (an expected average of 3 months)
  Antioxidative markers will be used to reflect the changes on oxidative stress. In particular, we will be analyzing the total antioxidant capacity (TAC).
Change scores of Glucose indicator | Baseline, posttest (an expected average of 3 months)
  HbA1C level will be tested to investigate the relationships between blood glucose level and aerobic exercise.
Change scores of Plasma lipid level | Baseline, posttest (an expected average of 3 months)
  The cholesterol ratio (total cholesterol divided by high-density lipid) will be evaluated to reflect the lipid level in the blood.
Change scores of Functional Independence Measure (FIM) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Lawton Instrumental Activities of Daily Living Scale (Lawton IADL) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Stroke Impact Scale (SIS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Caregiver Burden (CB) scale | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of EuroQol (EQ)-5D questionnaire | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Timed up and go test (TUG) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Six-minute walk test (6MWT) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Mobility level | Baseline, posttest (an expected average of 3 months)
Change scores of International Physical Activity Questionnaires (IPAQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Fugl-Meyer Assessment (FMA) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Rivermead Mobility Index (RMI) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of muscle strength | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
  We will evaluate isometric knee flexors and extensors muscle strength using handheld dynamometer. Also, we will use hand dynamometer to measure grip strength of the affected and less affected hand while the participant is seated, with the elbow at 90-degree flexion. We will record the mean value of 3 attempts.
Change scores of Community Integration Questionnaire (CIQ) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Change scores of Geriatric Depression Scale (GDS) | Baseline, posttest (an expected average of 3 months), follow-up (up to 9 months)
Genotyping of the BDNF val66met polymorphism | Between baseline and posttest (an expected average of 3 months)

CONTACTS AND LOCATIONS:
Locations (6):
- Taiwan (6):
  - Chang Gung Memorial Hospital, Kwei-Shan, Taoyuan
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Keeling Chang Gung Memorial Hospital, Keelung
  - Taipei Chang Gung Memorial Hospital, Taipei
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan

REFERENCES:
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186
- [Derived] Yeh TT, Wu CY, Hsieh YW, Chang KC, Lee LC, Hung JW, Lin KC, Teng CH, Liao YH. Synergistic effects of aerobic exercise and cognitive training on cognition, physiological markers, daily function, and quality of life in stroke survivors with cognitive decline: study protocol for a randomized controlled trial. Trials. 2017 Aug 31;18(1):405. doi: 10.1186/s13063-017-2153-7. PMID 28859664